CLINICAL TRIAL: NCT03039478
Title: Effect of Different Concentrations of Xylitol and Erythritol on the Release of Gastrointestinal Peptides and on Gastric Emptying Rates in Healthy Normal Weight Humans
Brief Title: Effect of Different Concentrations of Xylitol and Erythritol on Gut Peptide Release and Gastric Emptying in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PolyDose
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Physiological Satiation Mechanisms
MeSH Terms: interventions — Xylitol; Erythritol

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Xylitol 7g in 300mL tap water (Active Comparator): 12 volunteers receive 7g xylitol in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Xylitol 7g
- Xylitol 17g in 300mL tap water (Active Comparator): 12 volunteers receive 17g xylitol in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Xylitol 17g
- Xylitol 35g in 300mL tap water (Active Comparator): 12 volunteers receive 35g xylitol in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Xylitol 35g
- Erythritol 10g in 300mL tap water (Active Comparator): 12 volunteers receive 10g erythritol in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Erythritol 10g
- Erythritol 25g in 300mL tap water (Active Comparator): 12 volunteers receive 25g erythritol in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Erythritol 25g
- Erythritol 50g in 300mL tap water (Active Comparator): 12 volunteers receive 50g erythritol in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Erythritol 50g

INTERVENTIONS:
Dietary Supplement: Xylitol 7g — Xylitol 7g in 300mL tap water
  Other Names: E967-Xylitol
  Arms: Xylitol 7g in 300mL tap water
Dietary Supplement: Erythritol 10g — Erythritol 10g in 300mL tap water
  Other Names: E968-Erythritol
  Arms: Erythritol 10g in 300mL tap water
Dietary Supplement: Xylitol 17g — Xylitol 17g in 300mL tap water
  Other Names: E967-Xylitol
  Arms: Xylitol 17g in 300mL tap water
Dietary Supplement: Xylitol 35g — Xylitol 35g in 300mL tap water
  Other Names: E967-Xylitol
  Arms: Xylitol 35g in 300mL tap water
Dietary Supplement: Erythritol 25g — Erythritol 25g in 300mL tap water
  Other Names: E968-Erythritol
  Arms: Erythritol 25g in 300mL tap water
Dietary Supplement: Erythritol 50g — Erythritol 50g in 300mL tap water
  Other Names: E968-Erythritol
  Arms: Erythritol 50g in 300mL tap water

SUMMARY:
Xylitol and erythritol have become increasingly popular as sugar substitutes in the food industry. Both substances are freely available. While glucose ingestion stimulates satiation hormone secretion in the gut and slows down gastric emptying, artificial sweeteners such as aspartame, sucralose and acesulfame-K have no such effect. However, acute intake of 50g xylitol or 75g erythritol in 300mL tap water leads to a marked increase in the satiation hormones and induces a significant retardation in gastric emptying. The concentrations used to Show this effect were rather high (50g xylitol and 75g erythritol) and led to bloating and diarrhea in 60-70% of all subjects two hours after administration. The aim of the present study is to find an effective concentration of xylitol and erythritol still stimulating satiation hormone release without any gastrointestinal adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight subjects with a body-mass index of 19.0-24.9
* Normal eating habits (no diets; no dietary changes; no special dietary habits, such as vegetarian/vegan)
* Age 18-40 years
* Stable body weight for at least three months
* Informed Consent as documented by signature

Exclusion Criteria:

* Pre-existing consumption of xylitol or erythritol on a regular basis (usage of xylitol or erythritol as sugar replacement; xylitol or erythritol containing toothpaste is allowed)
* Regular intake of medications (except for oral contraceptives)
* Evidence of relevant cardiovascular, pulmonary, renal, hepatic, pancreatic, gastrointestinal, metabolic, endocrinological, neurological, psychiatric or other diseases at screening
* Clinically relevant abnormalities in haematological laboratory parameters
* Food allergies, food intolerance
* Pregnancy
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Acute effect on cholecystokinin ( CCK) release | changes from baseline to three hours after treatment
  effect on CCK release measured by a commercially available ELISA kit (enzyme-linked immunosorbent assay)

SECONDARY OUTCOMES:
Acute effects on gastric emptying | changes from baseline to three hours after treatment
  Acute effects on gastric emptying measured by 13C-sodium-acetate breath test
Acute effects on subjective feelings of hunger and satiety | changes from baseline to three hours after treatment
  Acute effects on subjective feelings of hunger and satiety measured by visual analogue scales

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided